CLINICAL TRIAL: NCT02486822
Title: The Management of Spontaneous Labour in Primigravida (SLiP): Labor Scale Versus WHO Partograph
Brief Title: Labor Scale Versus WHO Partograph in the Management of Labor
Acronym: SLiP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, M.B.B.Ch, M.S.c, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00008718 - SLiP
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Dystocia
Keywords: Labor scale; Partograph; Spontaneous labor; Primigravida
MeSH Terms: conditions — Dystocia | interventions — Amniotomy; Oxytocin; Cesarean Section

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Labor scale (Experimental): Observation Amniotomy Oxytocin Cesarean Section (CS)
  Interventions: Procedure: Amniotomy; Drug: Oxytocin; Procedure: Cesarean Section
- WHO partograph (Active Comparator): Observation Amniotomy Oxytocin Cesarean Section (CS)
  Interventions: Procedure: Amniotomy; Drug: Oxytocin; Procedure: Cesarean Section

INTERVENTIONS:
Procedure: Amniotomy — Amniotomy, artificial rupture of membranes, is done with initial delay of labor (in partograph: extension beyond alert line, in labor scale: when progress reaches the membrane line)
  Other Names: Artificial rupture of membranes
Drug: Oxytocin — Oxytocin augmentation: given with further delay of labour (according to the point of intervention of the partograph or the scale)
  Other Names: augmentation of labor
Procedure: Cesarean Section — Cesarean section: done when progress is deemed arrested (according to the definition of the partograph or the scale)
  Other Names: CS

SUMMARY:
This study aims to compare the novel labour scale with the traditional WHO partograph in the management of spontaneous labour in primigravida in terms of maternal and neonatal outcomes

DETAILED DESCRIPTION:
After many centuries through which vaginal delivery (VD) had been the only safe route of birth, Cesarean section (CS) emerged as an alternative in emergency situations. CS has gradually become an appealing option for both the mother and the obstetrician and its indications increase while CS was proving safety; the rate of CS in U.S.A increased by about 50% within 10 years around the beginning of the current century. However, the increasing prevalence of CS raises questions about the impact of this trend on maternal morbidity, mortality as well as its economic burden. Accordingly, recent guidelines have been directed to revise practice-base CS indications to only situations when CS is truly beneficial to the mother and/or the fetus.

Of these indications, the most reported one was labour dystocia. The WHO partograph is a famous chart that is commonly used to observe uncomplicated labour and is almost an objective approach to guide interference. Unfortunately, the rule of the partograph in reducing the incidence of CS is questionable. Furthermore, the design of the partograph is not exactly perfect to present the process of labour. For these reasons, the labour scale was designed as a novel follow-up chart during labour. The chart considered more objective and timed management of labour with more flexible range of time based on recent evidence. A previous pilot study on 77 women suggested that the labour scale may be a good alternative to the current partograph. This study is the first randomized trial the compares the 2 charts as regards the rate of CS, maternal and neonatal health outcomes and both patient and obstetrician satisfaction.

In this clinical trial, the investigators aim to compare the labour scale to the traditional WHO partograph in terms of incidence of labor dystocia and CS as well as maternal and neonatal outcomes

ELIGIBILITY:
Inclusion Criteria:

* Primigravida
* 38 - 42 weeks of gestation
* Singleton pregnancy
* Vertex presentation
* Spontaneous labour
* Average estimated fetal weight (2500 - 3800 gram)

Exclusion Criteria:

* Maternal medical or surgical major co-morbidity
* Previous uterine scar
* Induction of labor
* Premature rupture of membranes

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Successful vaginal delivery (reporting of whether labor ends in vaginal delivery or Cesarean Section. In case of CS, the indication will be reported) | Time of labor (maximum 24 hours)
  The proportion who delivered vaginal versus those indicated for Cesarean Section for labor dystocia

SECONDARY OUTCOMES:
Intrapartum maternal distress (assessed by clinical signs of maternal distress and dehydration) | Time of labor (maximum 24 hours)
Intrapartum maternal birth injuries (assessed clinically at the time of labor, the extent and type of repair and subsequent complications will be reported) | Time of labour and hospital stay (expected average 72 hours)
Primary postpartum hemorrhage evaluated by clinical signs, blood loss in mL, hemoglobin and interventions | The length of hospital stay (expected average 72 hours)
Maternal fever/postpartum infections as evaluated temperature, WBC count, CRP and culture | The length of hospital stay (expected average 72 hours)
Intrapartum fetal distress as diagnosed by fetal auscultation and electronic fetal monitoring | Duration of labor (maximum 24 hours)
birth injuries of the newborn (as reported by physical examination, documentation of birth injuries, and subsequent management ) | The length of hospital stay (expected average 1 week)
Neonatal distress "asphyxia" (as reported 1 & 5 minutes APGAR score, resuscitation event, umbilical artery pH, admission to NICU, length of stay and any further medical complications) | The length of hospital/NICU stay (expected average 1 week)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif AM Shazly, MBBCh,MSc, Principal Investigator — Assistant lecturer
Locations (1):
- Assiut Faculty of Medicine - Women Health Hospital, Asyut, Egypt

REFERENCES:
- [Background] Shazly SA, Embaby LH, Ali SS. The labour scale--assessment of the validity of a novel labour chart: a pilot study. Aust N Z J Obstet Gynaecol. 2014 Aug;54(4):322-6. doi: 10.1111/ajo.12209. Epub 2014 May 17. PMID 24835694
- [Background] Menacker F, Hamilton BE. Recent trends in cesarean delivery in the United States. NCHS Data Brief. 2010 Mar;(35):1-8. PMID 20334736
- [Background] Villar J, Valladares E, Wojdyla D, Zavaleta N, Carroli G, Velazco A, Shah A, Campodonico L, Bataglia V, Faundes A, Langer A, Narvaez A, Donner A, Romero M, Reynoso S, de Padua KS, Giordano D, Kublickas M, Acosta A; WHO 2005 global survey on maternal and perinatal health research group. Caesarean delivery rates and pregnancy outcomes: the 2005 WHO global survey on maternal and perinatal health in Latin America. Lancet. 2006 Jun 3;367(9525):1819-29. doi: 10.1016/S0140-6736(06)68704-7. PMID 16753484
- [Background] Liu S, Liston RM, Joseph KS, Heaman M, Sauve R, Kramer MS; Maternal Health Study Group of the Canadian Perinatal Surveillance System. Maternal mortality and severe morbidity associated with low-risk planned cesarean delivery versus planned vaginal delivery at term. CMAJ. 2007 Feb 13;176(4):455-60. doi: 10.1503/cmaj.060870. PMID 17296957
- [Background] Kjaergaard H, Olsen J, Ottesen B, Dykes AK. Incidence and outcomes of dystocia in the active phase of labor in term nulliparous women with spontaneous labor onset. Acta Obstet Gynecol Scand. 2009;88(4):402-7. doi: 10.1080/00016340902811001. PMID 19330572
- [Background] Gifford DS, Morton SC, Fiske M, Keesey J, Keeler E, Kahn KL. Lack of progress in labor as a reason for cesarean. Obstet Gynecol. 2000 Apr;95(4):589-95. doi: 10.1016/s0029-7844(99)00575-x. PMID 10725495
- [Background] Lavender T, Hart A, Smyth RM. Effect of partogram use on outcomes for women in spontaneous labour at term. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD005461. doi: 10.1002/14651858.CD005461.pub2. PMID 18843690
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Intrapartum Care: Care of Healthy Women and Their Babies During Childbirth. London: RCOG Press; 2007 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK49388/ PMID 21250397
- [Background] Amer-Wahlin I, Hellsten C, Noren H, Hagberg H, Herbst A, Kjellmer I, Lilja H, Lindoff C, Mansson M, Martensson L, Olofsson P, Sundstrom A, Marsal K. Cardiotocography only versus cardiotocography plus ST analysis of fetal electrocardiogram for intrapartum fetal monitoring: a Swedish randomised controlled trial. Lancet. 2001 Aug 18;358(9281):534-8. doi: 10.1016/s0140-6736(01)05703-8. PMID 11520523
- [Derived] Tolba SM, Ali SS, Mohammed AM, Michael AK, Abbas AM, Nassr AA, Shazly SA. Management of Spontaneous Labor in Primigravidae: Labor Scale versus WHO Partograph (SLiP Trial) Randomized Controlled Trial. Am J Perinatol. 2018 Jan;35(1):48-54. doi: 10.1055/s-0037-1605575. Epub 2017 Aug 8. PMID 28787749